CLINICAL TRIAL: NCT06409546
Title: Impact of Topical Pentoxifylline and Tocopherol in Treatment and Prevention of Medically-related Osteonecrosis of the Jaws: a Randomized Clinical Trial
Brief Title: Impact of Topical Pentoxifylline and Tocopherol in Treatment and Prevention of Medically-related Osteonecrosis of the Jaws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-31
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Medically Related Osteonecrosis of the Jaws
MeSH Terms: interventions — Tocopherols

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocopherol 75% and pentoxifilline 5% gel (Active Comparator): Patients treated with a topical gel of tocopherol 75% and pentoxifilline 5%
  Interventions: Drug: Tocopherol and pentoxifilline topical gel
- Placebo gel (Placebo Comparator): Patients treated with a topical placebo gel control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocopherol and pentoxifilline topical gel — Oral gel applied locally on the MRONJ related lesions or post-extraction sockets
  Arms: Tocopherol 75% and pentoxifilline 5% gel
Drug: Placebo — Oral gel applied locally on the MRONJ related lesions or post-extraction sockets
  Arms: Placebo gel

SUMMARY:
While there is no doubt about the benefits of antiresorptives, it is known that patients using these drugs are at increased risk of developing osteonecrosis of the jaws (MRNOJ), especially after oral procedures such as tooth extraction. The management of osteonecrosis has remained a controversial topic within the oral and maxillofacial surgery community.

The aim of the present study is to analyze the impact of topical pentoxifilline and tocopherol in the prevention and treatment of MRNOJ.

DETAILED DESCRIPTION:
A double-blind randomized controlled clinical trial is conducted in order to evaluate the impact of topical pentoxifilline and tocopherol in the prevention and treatment of MRNOJ and determine the statistical significance of the outcome variables.

48 subjects with MRNOJ, randomly allocated in two groups: placebo group with a 4% hydroxyethyl cellulose adhesive gel and the treatment group with the same gel containing pentoxifilline 5% and tocopherol 75%.

ELIGIBILITY:
Inclusion Criteria:

* Correspondence to the updated SIPMO criteria for MRONJ diagnosis
* Need for tooth extraction

Exclusion Criteria:

* Recent use of antibiotics and anti-inflammatories in the last 4 weeks
* Oral lesions of hard and soft tissues not related to MRONJ

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Oral Health Impact Profile Short Form (OHIP-14) | 6 months
  4-point scale in which the presence or absence of physical pain, functional limitation, psychological distress, physical, psychological and social disability and handicap is analyzed

SECONDARY OUTCOMES:
Alveolar bone resorption | 6 months
  Amount of vertical alveolar resorption expressed in mm

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Rodolico, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Pubmed
URL: https://pubmed.ncbi.nlm.nih.gov/